CLINICAL TRIAL: NCT02066740
Title: EverFlex™ Self-expanding Peripheral Stent With Entrust™ Delivery System Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP1007
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Diseases
Keywords: Superficial Femoral Artery; Proximal Popliteal Artery; Everflex; Entrust; stent
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EverFlex™ stent with Entrust™ delivery system (Experimental)
  Interventions: Device: EverFlex™ stent with Entrust™ delivery system

INTERVENTIONS:
Device: EverFlex™ stent with Entrust™ delivery system

SUMMARY:
The purpose of this study is to collect acute confirmatory data to evaluate technical success and acute safety of the EverFlex™ self-expanding peripheral stent with Entrust™ delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Has stenotic, restenotic (from PTA or adjunct therapy, not including stents or stent grafts),
* or occluded lesion(s) located in the superficial femoral artery (SFA) and/or proximal popliteal artery (PPA) suitable for primary stenting.

Exclusion Criteria:

* Has undergone previous implantation of stent(s) or stent graft(s) in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl M Wahlgren, MD/PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Klinikum Weiden, Weiden, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- EverFlex™ Stent With Entrust™ Delivery System: Subjects were treated with the EverFlex™ stent with Entrust™ delivery system
Period: Overall Study
Arm/Group | EverFlex™ Stent With Entrust™ Delivery System
Started | 34
Completed | 32
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- EverFlex™ Stent With Entrust™ Delivery System: EverFlex™ stent with Entrust™ delivery system
Arm/Group | EverFlex™ Stent With Entrust™ Delivery System
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Region of Enrollment [Number; unit: participants]
  Germany | 27
  Sweden | 7

OUTCOME MEASURES:

1. Primary Outcome: Absence of Stent Elongation
Description: Absence of stent elongation is achieved when the implanted stent length does not exceed the allowed stent length
Time Frame: Intra operative
Measure: Number; unit: percentage absence of stent elongation
Units Other Than Participants: Number of Stents Implanted
Arm/Group | EverFlex™ Stent With Entrust™ Delivery System
Number analyzed (Participants) | 34
Number analyzed (Number of Stents Implanted) | 45
percentage absence of stent elongation | 95.6

2. Primary Outcome: Successful Stent Deployment
Description: Successful stent deployment to be assessed based on stent delivery, lesion coverage and accuracy of deployment.
Time Frame: Procedure
Measure: Number; unit: percentage - successful stent deployment
Units Other Than Participants: Stents Implanted
Arm/Group | EverFlex™ Stent With Entrust™ Delivery System
Number analyzed (Participants) | 34
Number analyzed (Stents Implanted) | 45
percentage - successful stent deployment | 100.0

ADVERSE EVENTS:
Description: Only procedure-related AEs, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects, and Unanticipated Serious Adverse Device Effects were required to be reported.
Arm/Group | EverFlex™ Stent With Entrust™ Delivery System
Serious Adverse Events (participants affected / at risk) | 4/34
Other Adverse Events (participants affected / at risk) | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EverFlex™ Stent With Entrust™ Delivery System (N=34)
Gastronintestinal disorders (Gastrointestinal disorders) | 1 (1)
General disorders (General disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (2)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)
Vascular disorders (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and Sponsor [or its agents] that restricts PI's rights to discuss or publish trial results without permission of the Sponsor.

Trial is still ongoing.